CLINICAL TRIAL: NCT06619652
Title: Knowledge of Egyptian Dental Practitioners Regarding Diagnosis and Management of Root Caries: a Cross-sectional Study
Brief Title: Egyptian Dentists Knowledge Regarding the Diagnosis and Management of Root Caries
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Gamal Abdel-Hakim, principle investigator, Cairo University
Other Study IDs: 14422022412792
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Root Caries
Keywords: root caries; knowledge
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a cross-sectional study that aims to assess the knowledge of a sample of Egyptian dental practitioners regarding the diagnosis and management of root caries Dental caries is a major problem for adults in both developing and industrialized countries. As individuals get older, the prevalence of caries tends to increase.In recent decades, life expectancy has been steadily increasing. A report published by the United Nations in 2020 states that the global population of people aged 65 and over is currently 703 million, and it is expected to double in thirty years.However, this increase in life expectancy has led to an increase in health issues among the elderly, including the risk of developing root caries lesions. Root caries develop when the root surface is exposed to the oral cavity due to loss of alveolar bone height and subsequent gingival recession, leading to the softening of the tooth structure.

This lesion presents a complex challenge for dental practitioners. Surgical intervention is difficult due to moisture contamination and the lesions proximity to the pulp chamber. Accurately assessing the risk and implementing appropriate preventive strategies can reduce the need for complex restorative treatments and associated dental problems

DETAILED DESCRIPTION:
Recently, there has been growing concern about root caries lesions in routine dental practice.The concern regarding this condition is increasing, mainly linked to the discrepancies in how dentists manage root caries.Diagnosing root caries can be challenging due to limited visibility, and it requires careful examination without forceful probing of the tissue. Furthermore, the successful management of root carious lesions can be affected by various factors, including the operator expertise, knowledge, and the chosen treatment approach.

These factors shape the decisions they make in their practice, including the selection of restorative materials and operative techniques.Thus, every effort needs to be made to better understand the current state of practice and trends relating to root caries management which will be of benefit to dentists universally in the practice of dentistry.

Understanding dentist knowledge about root caries is highly important as they play a central role in the prevention, early detection and appropriate treatment of root caries.Gaps or deficiencies in their diagnostic skills or treatment decision-making could lead to missed or delayed diagnosis, suboptimal treatment and poor outcome for the patients By identifying areas where dentists may lack sufficient knowledge in managing root caries, the findings of this study can guide updates to dental school curricula and clinical practice guidelines. strengthening dentist competence in diagnosing and managing root caries will ultimately improve the quality of care delivered to the patients

Aim of the study:

The aim of this study is to assess the knowledge of Egyptian dental practitioners regarding diagnosis and management of root caries

Research question:

What is the knowledge of a sample of Egyptian dental practitioners about diagnosis and management of root caries lesions?

POTS:

Population: A sample of Egyptian dental practitioner Primary outcome: knowledge about diagnosis and management of root caries lesion Time: academic year 2024-2025 Study design: cross-sectional.

Methods:

Study design:

Observational cross-sectional study on a sample of Egyptian dental practitioners.

Settings:

The study is a cross-sectional study utilizing an electronic self-administered questionnaire (SAQ) assessing the knowledge of Egyptian dental practitioners regarding the diagnosis and management of root caries.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian dental practitioners that have completed their bachelor's degree, have practice license and registered in the Egyptian Dental Syndicate.

Exclusion Criteria:

* Undergraduate dental students
* Dental interns

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sample of Egyptian dental practitioners
Sampling Method: Probability Sample
Enrollment: 355 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Egyptian dentists | 1 year
  Dentist knowledge about the diagnosis and management of root caries by survey questionnaire the questionnaire consists of 3 categories Category1: General clinical routine Category2: Knowledge and practices related to two clinical cases Category3: Participants demographics

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided